CLINICAL TRIAL: NCT01410435
Title: An Open-label, Multi-Centre, Non-Randomised Extension Study to Assess the Ability to Maintain a Stable Haemoglobin and to Assess Safety of Iron Isomaltoside 1000 (Monofer®) in Subjects With Inflammatory Bowel Disease
Brief Title: Safety and Efficacy Extension Study of Iron Isomaltoside 1000 (Monofer®) in Subjects With Inflammatory Bowel Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-IBD-01-Extension
Record Dates: First submitted 2011-07-06; First posted 2011-08-05 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Inflammatory Bowel Disease; Anaemia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Monofer

INTERVENTIONS:
Drug: Monofer — Infusion according to current HB level

SUMMARY:
Since the duration of most studies with IV iron in IBD subjects have been only 4-12 weeks studies there is a need to follow-up on long term safety and efficacy of any maintenance iron therapy.

This study represents subjects from the Lead-in Study (P-Monofer-IBD-01) on iron isomaltoside 1000 (Monofer®) to assess the long term safety of iron isomaltoside 1000 (Monofer®) and its ability to maintain stable haemoglobin in IBD subjects with Iron Deficiency Anaemia (IDA).

ELIGIBILITY:
Inclusion Criteria:

1. Completed the Lead-in Study or discontinued from Lead-in Study due to intolerance to oral iron.
2. Life expectancy beyond 18 months by Investigator's judgement.
3. Willingness to participate after informed consent. -

Exclusion Criteria:

1. Discontinuation from Lead-in Study (except for due to intolerance to oral therapy).
2. Any major protocol deviation in Lead-in Study.
3. Pregnancy and nursing [To avoid pregnancy, women have to be postmenopausal, surgically sterile, or women of child bearing potential must use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product (5 days): Contraceptive pills, Intrauterine Devices (IUD), contraceptive injections (prolonged-release gestagen), subdermal implantation, vaginal ring, and transdermal patches].
4. Any other medical condition that, in the opinion of Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study.
5. Patients with a Harvey-Bradshaw Index >8 or Partial Mayo Score (excluding Endoscopy Sub-score) >6 at End of Study Visit of Lead-in Study.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Long term efficacy | Baseline to month 12
  1. To assess the long term efficacy of iron isomaltoside 1000 (Monofer®) by means of the ability to maintain stable Hb (defined as Hb ≥ 12.0 g/dL) in subjects with Hb ≥ 12.0 g/dL at the Baseline of Extension Study.
  2. To assess the ability to achieve stable Hb (Hb ≥ 12.0 g/dL) at Month 3 Visit of Extension Study, and then to maintain the stable Hb thereafter in subjects with Hb < 12.0 g/dL at Baseline of Extension Study.

SECONDARY OUTCOMES:
Long term safety | Baseline to month 12
  To assess the long term safety of iron isomaltoside 1000 (Monofer®) maintenance, measured through laboratory testings and number of subjects who experience any adverse drug reaction.

CONTACTS AND LOCATIONS:
Locations (2):
- Austria, Austria, Austria
- Hungary, Hungary, Hungary